CLINICAL TRIAL: NCT02101086
Title: Evaluation of the Efficacy and Safety of Autologous Cord Blood Transfusions in Premature Infants
Brief Title: Autologous Cord Blood Transfusion in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emel Okulu, MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ankara University-06
Record Dates: First submitted 2014-03-28; First posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Anemia of Prematurity
Keywords: umbilical cord blood; premature; autologous transfusion; allogeneic transfusion
MeSH Terms: conditions — Anemia; Premature Birth | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Cord Blood Transfusion (Experimental): Autologous cord blood transfusion 10 mL per kg for anemia
  Interventions: Other: Blood transfusion
- Allogeneic blood transfusion (Active Comparator): Allogeneic blood transfusion 10 mL per kg for anemia
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Whenever the infant indicated to receive transfusion, a blood product request was sent to the blood bank. This infant was randomly assigned to the autologous or the allogeneic product labeled for each patient at birth in the blood bank

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous cord blood transfusions in very-low-birth-weight premature infants, and to evaluate the developmental outcomes of the infants who received autologous transfusions.

DETAILED DESCRIPTION:
Blood transfusions have many risks including transfusion reactions and infections. Cord blood is accepted as an alternative method for red cell transfusions in low-birth weight (LBW) premature newborns. However, experience and scientific evidence concerning in-vivo efficacy and safety of red blood cell (RBC) concentrates derived from cord blood in very LBW premature newborns is still insufficient.

A total of 50 umbilical cord blood (UCB) collected from infants born before 32 weeks' gestational age and processed into autologous RBC products. Infants requiring blood transfusion were randomly assigned to an autologous or allogeneic product. Two randomized groups were compared on the 14th, 28th, 35th days and >35th days with respect to hemoglobin levels, transfusion numbers, transfusion and phlebotomy volumes, and hemoglobin, reticulocyte counts and erythropoietin levels in the postconceptional 36th and 40th weeks' gestation, and hemoglobin levels at postnatal 6-months age. All transfused infants were developmentally assessed by the end of the postnatal first year.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at ≤ 32 weeks gestational age
* Parental consent

Exclusion Criteria:

* rhesus incompatibility
* hydrops fetalis
* maternal viral or bacterial infections including suspected chorioamnionitis
* parental refuse

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants that receive autologous transfusion with a decrease in allogeneic transfusion | one year

SECONDARY OUTCOMES:
The hemoglobin levels at postnatal 14th days | 14 days
The hemoglobin levels at postnatal 28th days | 28 days
The hemoglobin levels at postnatal 35th days | 35 days
The hemoglobin, erythropoietin and reticulocyte counts at postconceptional 36 weeks | 3 months
The hemoglobin, erythropoietin and reticulocyte counts at postconceptional 40 weeks | 5 months
Developmental assessments of infants | One year

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Arsan, Professor, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)